CLINICAL TRIAL: NCT00057837
Title: A Randomized Phase II Study: Sequencing Topoisomerase Inhibitors for Extensive Stage Small Cell Lung Cancer (SCLC): Topotecan Sequenced With Etoposide/Cisplatin, and Irinotecan/Cisplatin Sequenced With Etoposide
Brief Title: Comparison of Two Combination Chemotherapy Regimens in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000276590; U10CA021115 (NIH); E5501 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: extensive stage small cell lung cancer; Topotecan; Etoposide; Cisplatin; Irinotecan
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Cisplatin; Platinum; Etoposide; Podophyllotoxin; Irinotecan; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET (Topotecan/Etoposide/Cisplatin/G-CSF) (Experimental): Patients receive topotecan intravenously (IV) over 30 minutes on days 1-3; etoposide IV over 60 minutes immediately followed by cisplatin IV over 60 minutes on days 8-10; and filgrastim (G-CSF) subcutaneously daily beginning on day 11 and continuing until blood counts recover.
  Interventions: Biological: G-CSF; Drug: Cisplatin; Drug: Etoposide; Drug: Topotecan
- PIE (Irinotecan/Cisplatin/Etoposide) (Experimental): Patients receive irinotecan IV over 90 minutes and cisplatin IV over 60 minutes on days 1 and 8 and oral etoposide twice daily on days 3 and 10 of each cycle.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Irinotecan

INTERVENTIONS:
Biological: G-CSF — G-CSF will be administered subcutaneously at a dose of 5 mcg/kg once a day starting on day 11 until WBC recovery > 10,000 dL.
  Other Names: Filgrastim; Neupogen; recombinant-rnethionyl human granulocyte-colony stimulating factor; granulocyte colony-stimulating factor; r-metHuG-CSF
  Arms: PET (Topotecan/Etoposide/Cisplatin/G-CSF)
Drug: Cisplatin — Arm PET: 20 mg/m2 IV on days 8, 9 and 10 of each cycle following Etoposide. Arm PIE: 20 mg/m2 IV on days 1 and 8 of each cycle following Irinotecan.
  Other Names: Platinol®; Cis-diaminedichloroplatinum; Cis-diaminedichloroplatinum (II); diaminedichloroplatinum; cis-platinum; platinum; Platinol; Platinol-AQ; DDP; CDDP; DACP; NSC 119875
Drug: Etoposide — Arm PET: 70 mg/m2 IV over 60 minutes on days 8, 9 and 10 of each cycle. Arm PIE: 85 mg/m2 orally (divided into 2 doses, 12 hours apart) on day 3 and 10 of each cycle.
  Other Names: VP-16; VePesid; VP-16-213; EPEG; epipodophyllotoxin; NSC # 141540
Drug: Irinotecan — 50 mg/m2 IV over 90 minutes on days 1 and 8 of each cycle (Arm PIE only).
  Other Names: Camptothecin-11; CPT-11
  Arms: PIE (Irinotecan/Cisplatin/Etoposide)
Drug: Topotecan — Topotecan 0.75 mg/m2 IV over 30 minutes on days 1,2 and 3 of each cycle (Arm PET only).
  Other Names: Hycamtin®; Hycamptamine; SK&F 104864-A; Topotecan Formula AS
  Arms: PET (Topotecan/Etoposide/Cisplatin/G-CSF)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating extensive-stage small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the response frequency of patients with extensive stage small cell lung cancer treated with topotecan, cisplatin, and etoposide and with irinotecan, cisplatin, and etoposide.
* Evaluate the toxic effects of these regimens in these patients.
* Evaluate the duration of response and survival of patients treated with these regimens.

Secondary

* To investigate the occurrence of various breast cancer resistance protein (BCRP) alleles in patients receiving topoisomerase 1 inhibitors and their impact on clinical response and toxicity.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (PET): Patients receive topotecan intravenously (IV) over 30 minutes on days 1-3; etoposide IV over 60 minutes immediately followed by cisplatin IV over 60 minutes on days 8-10; and filgrastim (G-CSF) subcutaneously daily beginning on day 11 and continuing until blood counts recover.
* Arm II (PIE): Patients receive irinotecan IV over 90 minutes and cisplatin IV over 60 minutes on days 1 and 8 and oral etoposide twice daily on days 3 and 10.

In both arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ACTUAL ACCRUAL: A total of 140 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Extensive stage small cell lung cancer (SCLC) with measurable disease, evaluated within 2 weeks prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Disease-free for >=5 years if had a prior second malignancy other than treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
* Adequate hematologic, hepatic and renal function determined by the following tests, within 4 weeks prior to randomization: white blood cell (WBC) >=4000/mm3 and platelets >=100,000/mm3; bilirubin <= upper limit of normal; serum glutamic pyruvate transaminase (SGPT) or alanine transaminase (ALT) and serum glutamic oxaloacetic transaminase (SGOT) or aspartate transaminase( AST) <=2.5 x upper limit of normal if no demonstrable liver metastases or <=5 times upper limit of normal in the presence of liver metastases; Calculated creatinine clearance >=30 using the formulas in the protocol
* Age 18 and older
* Strongly advised to use an accepted and effective method of contraception
* Those with central nervous system (CNS) metastases were eligible if the metastases were treated without advancing symptoms prior to the initiation of chemotherapy
* Those receiving erythropoietin could continue to receive it

EXCLUSION CRITERIA:

* Prior radiotherapy for lung cancer; Prior radiotherapy allowed only for central nervous system (CNS) metastases
* Prior chemotherapy for this disease
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-07-14 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Aisner, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (79):
- United States (79):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Hematology & Oncology Care, Moline, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Bettendorf, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Regional Cancer Center at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on March 24, 2004, accrued its first patient on July 14, 2004, and was closed on April 14, 2008 with final accrual of 140 patients.
Period: Overall Study
Arm/Group | PET (Topotecan/Etoposide/Cisplatin/G-CSF) | PIE (Irinotecan/Cisplatin/Etoposide)
Started | 70 | 70
Treated | 69 | 68
Eligible and Treated | 66 | 66
Patients With Response | 46 | 38
Completed | 39 | 31
Not Completed | 31 | 39
Not completed — Progression/relapse | 12 | 14
Not completed — Adverse Event | 2 | 12
Not completed — Death | 5 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Alternative therapy | 0 | 1
Not completed — Other complicating disease | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Ineligible | 3 | 3
Not completed — Never started treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PET (Topotecan/Etoposide/Cisplatin/G-CSF) | PIE (Irinotecan/Cisplatin/Etoposide) | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 76] | 64 [44 to 83] | 63 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 33 | 58
  Male | 41 | 33 | 74

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Response by Solid Tumor Response Criteria (RECIST)
Description: Per RECIST criteria, Complete response (CR)= disappearance of all target and nontarget lesions Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
  Objective response = CR + PR
Time Frame: Assessed every 6 weeks while on treatment, and then every 3 months for patients < 2 years from study entry, every 6 months if patient is 2-3 years from study entry.
Population: Only treated and eligible patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | PET (Topotecan/Etoposide/Cisplatin/G-CSF) | PIE (Irinotecan/Cisplatin/Etoposide)
Number analyzed (Participants) | 66 | 66
proportion of participants | 0.697 [0.591 to 0.789] | 0.576 [0.467 to 0.679]

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented, taking as reference the smallest measurements recorded since treatment started.
Time Frame: as for outcome 1
Population: Only eligible and treated patients with response are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PET (Topotecan/Etoposide/Cisplatin/G-CSF) | PIE (Irinotecan/Cisplatin/Etoposide)
Number analyzed (Participants) | 46 | 38
Months | 6.0 [5.0 to 7.0] | 6.0 [5.0 to 8.3]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 1 years
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PET (Topotecan/Etoposide/Cisplatin/G-CSF) | PIE (Irinotecan/Cisplatin/Etoposide)
Number analyzed (Participants) | 66 | 66
Months | 11.9 [9.6 to 13.7] | 11.0 [8.6 to 13.1]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | PET (Topotecan/Etoposide/Cisplatin/G-CSF) | PIE (Irinotecan/Cisplatin/Etoposide)
Serious Adverse Events (participants affected / at risk) | 48/69 | 51/68
Other Adverse Events (participants affected / at risk) | 66/69 | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET (Topotecan/Etoposide/Cisplatin/G-CSF) (N=69) | PIE (Irinotecan/Cisplatin/Etoposide) (N=68)
Anemia (Blood and lymphatic system disorders) | 14 | 5
Leukopenia (Investigations) | 13 | 22
Neutropenia (Investigations) | 23 | 31
Thrombocytopenia (Investigations) | 15 | 3
Transfusion: Platelets (Investigations) | 1 | 0
Transfusion: PRBCS (Injury, poisoning and procedural complications) | 18 | 11
Supraventricular arrhythmias (Cardiac disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Thrombosis/Embolism (Vascular disorders) | 0 | 1
Visceral Arterial Ischemia (Vascular disorders) | 1 | 0
Cardiac-other (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 10 | 11
Weight loss (Investigations) | 1 | 1
Constitutional symptoms (Investigations) | 0 | 1
Skin- Other (Skin and subcutaneous tissue disorders) | 0 | 1
SIADH (The syndrome of inappropriate antidiuretic hormone secretion) (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2 | 17
GI-other (Gastrointestinal disorders) | 0 | 1
Hemorrhage with Grade 3 or 4 Platelets (Vascular disorders) | 0 | 1
CNS hemorrhage (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1
Bilirubin increased (Investigations) | 1 | 1
AST increased (Investigations) | 2 | 1
ALT increased (Investigations) | 3 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Infection w/ Gr3-4 neutropenia (Infections and infestations) | 4 | 5
Infection w/ unknown ANC (Infections and infestations) | 1 | 1
Infection w/o neutropenia (Infections and infestations) | 3 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Confusion (Psychiatric disorders) | 0 | 2
Depressed level of consciousness (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Earache (Ear and labyrinth disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary- Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PET (Topotecan/Etoposide/Cisplatin/G-CSF) (N=69) | PIE (Irinotecan/Cisplatin/Etoposide) (N=68)
Anemia (Blood and lymphatic system disorders) | 65 | 64
Leukopenia (Investigations) | 53 | 59
Lymphopenia (Investigations) | 1 | 5
Neutropenia (Investigations) | 47 | 56
Thrombocytopenia (Investigations) | 46 | 34
Edema (General disorders) | 4 | 7
Hypotension (Vascular disorders) | 6 | 6
Fatigue (General disorders) | 50 | 53
Fever (General disorders) | 7 | 6
Rigors/chills (General disorders) | 1 | 4
Weight gain (Investigations) | 5 | 4
Weight loss (Investigations) | 14 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 33
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 5
Anorexia (Metabolism and nutrition disorders) | 22 | 32
Constipation (Gastrointestinal disorders) | 18 | 15
Dehydration (Metabolism and nutrition disorders) | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 4 | 7
Dry mouth (Gastrointestinal disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 42 | 49
Stomatitis (Gastrointestinal disorders) | 14 | 10
Taste disturbance (Nervous system disorders) | 11 | 11
Vomiting (Gastrointestinal disorders) | 16 | 22
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 12 | 34
Alkaline phosphatase increased (Investigations) | 37 | 22
Bilirubin increased (Investigations) | 7 | 6
AST increased (Investigations) | 14 | 16
ALT increased (Investigations) | 19 | 18
Infection w/o neutropenia (Infections and infestations) | 8 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 28 | 34
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 | 4
Dizziness/Lightheadedness (Nervous system disorders) | 8 | 10
Insomnia (Psychiatric disorders) | 5 | 7
Depression (Psychiatric disorders) | 3 | 5
Neuropathy-sensory (Nervous system disorders) | 12 | 13
Abdominal Pain (Gastrointestinal disorders) | 1 | 7
Bone, pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Creatinine increased (Investigations) | 15 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No